CLINICAL TRIAL: NCT05690217
Title: The Difference in the Biological Characteristic Characteristics of the Heart and Lung Meridians Between COPD Patients and Healthy Subjects
Brief Title: The Difference in the Biological Characteristic Characteristics of the Heart and Lung Meridians
Status: Completed | Type: Observational
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Hantong Hu, Attending doctor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Other Study IDs: ZSLL-KY-2019-001
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: acupuncture; meridians; biological characteristic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD group: There are 40 chronic obstructive pulmonary disease (COPD) patients in the COPD group.
- Healthy control group: There are 40 age-matched healthy participants in the healthy control group.

SUMMARY:
The association between viscera and the body surface remains obscure, but a better understanding of it will maximize its diagnostic and therapeutic values in clinical practice. Therefore, this study aimed to investigate the specificity of the association between viscera and the body surface in the pathological state.

DETAILED DESCRIPTION:
Study subjects included 40 chronic obstructive pulmonary disease (COPD) participants in the COPD group and 40 age-matched healthy participants in the healthy control group. Laser doppler flowmetry, infrared thermography, and functional near-infrared spectroscopy were respectively adopted to measure (1) the perfusion unit (PU), (2) temperature, and (3) regional oxygen saturation (rSO2) of 4 specific somatic sites distributing in the heart and lung meridians. These 3 outcome measures reflected the microcirculatory, thermal and metabolic characteristics of the body surface, respectively.

ELIGIBILITY:
Inclusion Criteria:

* COPD participants were eligible if they 1) satisfied the diagnostic criteria of COPD; 2) were in the stable phase of COPD; 3) were 20 ≤ age ≤ 75 years; 4) fully understood the study protocol and signed the written informed consent. Healthy participants were eligible if they 1) were healthy subjects who provided a medical examination report within 6 preceding months for confirming their health conditions; 2) were age-matched with the COPD group; 3) fully understood the study protocol and signed the written informed consent.

Exclusion Criteria:

* COPD patients were excluded if they 1) had other major lung diseases, such as bronchiectasis, pneumothorax, and lung tumors; 2) had concomitant heart diseases; 3) had serious concomitant diseases in major systems that were not controlled effectively 4) had mental diseases, history of drug abuse, and alcohol dependence; 5) were lactating or pregnant and 6)had scarring, hyperpigmentation, redness, swelling and heat in the skin around the measurement sites, which would affect the accuracy of examinations. Healthy subjects were excluded if they 1) had mental illness, history of drug abuse and alcohol dependence; 2) were lactating or pregnant; 3) had scarring, hyperpigmentation, redness, swelling, and heat in the skin around the measurement sites, which would affect the accuracy of examinations.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The diagnostic criteria of COPD were based on criteria proposed by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) consensus published in 2017, in which persistent airflow obstruction is confirmed according to the pulmonary function test. Healthy participants were determined by a medical examination report within 6 preceding months for confirming their health conditions.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Perfusion unit | Baseline
  Perfusion unit of acupuncture points is measured by Laser doppler flowmetry
Temperature | Baseline
  Temperature of acupuncture points is measured by infrared thermography
Regional oxygen saturation | Baseline
  Regional oxygen saturation of acupuncture points is measured by functional near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No